CLINICAL TRIAL: NCT01470209
Title: A Phase I Study of BKM120 and Everolimus in Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Taofeek K. Owonikoko, Professor and Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00048549; WCI1925-10 (Other: Other)
Record Dates: First submitted 2011-10-25; First posted 2011-11-11 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Solid Tumors; Lung Cancer
Keywords: lung cancer with activated mTOR/PI3K pathway; alterations in PIK3CA, NF1, TSC1/TSC2, mTOR, KRAS, LKB1, PTEN
MeSH Terms: conditions — Lung Neoplasms; Hereditary Sensory and Autonomic Neuropathies | interventions — NVP-BKM120; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination of BKM120 and everolimus (Experimental)
  Interventions: Drug: BKM120; Drug: Everolimus

INTERVENTIONS:
Drug: BKM120 — BKM120 (20mg to 100mg) will be self-administered (by the patients themselves). The investigator will instruct the patient to take the study drug exactly as specified in the protocol. BKM120 will be administered on a continuous once daily dosing schedule. Patients should be instructed to take the dose of BKM120 daily in the morning, one hour after a light breakfast (morning meal) at approximately the same time each day. BKM120 should be taken with a glass of water and consumed over as short a time as possible. Patients should swallow the capsules as a whole and not chew them. Patients should continue to fast for 2 hours after the administration of each BKM120 dose.
  Other Names: Buparlisib
Drug: Everolimus — RAD001 will be self-administered (by the patients themselves). The investigator will instruct the patient to take the study drug exactly as specified in the protocol. RAD001 will be administered orally as once daily dose of 5mg or 10 mg (based on the dose cohort) continuously from study day 1 until progression of disease or unacceptable toxicity. Patients will be instructed to take RAD001 in the morning, at the same time each day.
  Other Names: RAD001; Afinitor

SUMMARY:
This study will assess the safety of combining two agents (everolimus and BKM120) for the treatment of advanced cancer arising from solid organ in patients who are no longer benefiting from or unable to withstand standard treatment of these conditions.

DETAILED DESCRIPTION:
The purpose of this study is to study the combination of two anticancer drugs, everolimus (RAD001) and BKM120, in patients whose cancer is no longer responding to standard treatment or patients who are unable to tolerate the standard treatment for their cancer. The investigators seek to establish the safety of taking these two medications together and to determine the appropriate doses of the two drugs when given together as well as identify potential side effects when the drugs are administered together.

Another purpose of this study is to determine the effectiveness and side effects of the combination of RAD001 and BKM120 by looking at the patient's response to the treatment. The investigators want to find out what effects, good or bad, the drugs have on the patient's cancer.

This study will also look at specific biomarkers in the patient's blood and in the tumor tissue which are involved in the growth of tumor cells and determine if the levels of these biomarkers are related to the patient's response to treatment or development of side effects.

Everolimus, also known by the brand name, Afinitor, is a biologic drug approved by the Food and Drug Administration (FDA) for the treatment of kidney cancer. It works by preventing cancer cell from multiplying and it also renders them easily susceptible to death.

BKM120 is a new study drug that is being tested for its ability to treat cancer. However, it has not yet been approved by the FDA for the treatment of any specific cancer type.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic confirmation of a solid malignancy with established intolerance or refractoriness to standard therapies
2. Age ≥ 18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
4. Patients must have at least one site of measurable disease (per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria)
5. Adequate organ function including:

   1. Bone marrow function as shown by: absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L, platelets ≥ 100 x 10⁹/L, Hb >9 g/dL
   2. Electrolytes: Total calcium (corrected for serum albumin) within normal limits (ongoing requirement for bisphosphonate to control malignant hypercalcemia is not allowed but prophylactic use of bisphosphonate to prevent skeletal complication of bone metastasis is allowed); magnesium ≥ the lower limit of normal
   3. Liver function: aspartate aminotransferase (AST)/serum glutamate oxaloacetate transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) ≤ 2.5 x Upper Limit of Normal (ULN) or ≤ 5.0 x ULN if liver metastases are present; serum bilirubin ≤ 1.5 x ULN in patients with known Gilbert Syndrome, total bilirubin ≤ 3 x ULN, with direct bilirubin ≤ 1.5 x ULN
   4. Renal function: serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 50 mL/min or calculated glomerular filtration rate (GFR) of 60cc/ml using the formula of Cockroft and Gault
6. Serum amylase ≤ ULN
7. Serum lipase ≤ ULN
8. Fasting plasma glucose ≤ 120 mg/dL (6.7 mmol/L)
9. International normalized ratio (INR) ≤ 2
10. Negative serum pregnancy test within 48 hours before starting study treatment in women with childbearing potential
11. Ability and willingness to participate in the informed consent process and signing a copy of the informed consent form
12. Presence of appropriate size and site of viable tumor tissue for safe tumor biopsy collection (the biopsy is optional and requirement is only applicable to subjects considered for the expansion cohort stage of the study)
13. Ability and willingness to undergo repeat tumor biopsies (the biopsy is optional and only applicable to subjects considered for the expansion cohort stage of the study)

Exclusion Criteria:

1. Patients who have received prior treatment with a phosphatidylinositol 3-kinase (P13K) inhibitor or RAD001 (if discontinued for toxicity)
2. Patients with a known hypersensitivity to BKM120, RAD001 (including other rapalogs) or their excipients
3. Patients with untreated symptomatic brain metastases are excluded. However, patients with metastatic central nervous system (CNS) tumors may participate in this trial, if the patient is > 4 weeks from therapy completion (including radiation and/or surgery), is clinically stable at the time of study entry and is not receiving corticosteroid therapy for the brain mets.
4. Patients with acute or chronic liver, renal disease or pancreatitis
5. Patients has any of the following mood disorders as judged by the Investigator or a Psychiatrist, or who meets the cut-off score of ≥ 12 the Patient Health Questionnaire-9 (PHQ-9) or a cut-off of ≥ 15 in the Generalized Anxiety Disorder-7 (GAD-7) mood scale, respectively, or selects a positive response of '1, 2, or 3' to questions number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9) :

   1. Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others) or patients with active severe personality disorders are not eligible. Note: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous 6 weeks prior to start of study drug.
   2. ≥ Common Toxicity Criteria for Adverse Effects (CTCAE) grade 3 anxiety
   3. Note: The psychiatric judgment overrules the mood assessment questionnaire result or the investigators judgment.
6. Patient has active cardiac disease including any of the following:

   * Left ventricular ejection fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
   * Corrected QT interval (QTc) > 480 msec on screening ECG (using the Fridericia's corrected QT interval [QTcF] formula)
   * Angina pectoris that requires the use of anti-anginal medication
   * Ventricular arrhythmias except for benign premature ventricular contractions
   * Supraventricular and nodal arrythmias requiring a pacemaker or not controlled with medication
   * Conduction abnormality requiring a pacemaker
   * Valvular disease with document compromise in cardiac function
   * Symptomatic pericarditis
7. Patient has a history of cardiac dysfunction including any of the following:

   * Myocardial infraction within the last 6 months, documented by persistent elevated cardiac enzymes or preexistent regional wall abnormalities on assessment of LVEF function
   * History of or documented congestive heart failure (New York Heart Association functional classification III-IV)
   * Documented cardiomyopathy
8. Active diarrhea ≥ CTCAE grade 2
9. Patients with clinical manifestation of uncontrolled diabetes mellitus (i.e. treated and/or with clinical signs) or steroid-induced diabetes mellitus
10. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection). Patients with unresolved diarrhea will be excluded as previously indicated.
11. Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., granulocyte-colony stimulating factor [G-CSF], granulocyte macrophage-colony-stimulating factor [GM-CSF]) ≤ 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued.
12. Patients who are currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug. Please refer to Table 5-2 or a list of prohibited QT prolonging drugs with risk of Torsades de Pointes.
13. Patients receiving chronic treatment with steroids or another immunosuppressive agent. Note: Topical applications (e.g. for rash), inhaled sprays (e.g. for obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed. Patients with previously treated brain metastases, who are on stable low dose corticosteroid treatment (e.g. dexamethasone 2 mg/day, prednisolone 10 mg/day) for at least 14 days before start of study treatment are eligible.
14. Patients who have received chemotherapy or targeted anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug or who have not recovered from side effects of such therapy
15. Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) ≤ 5 effective half lives prior to starting study drug or who have not recovered from side effects of such therapy
16. Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
17. Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
18. Patients who are currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant.
19. Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control. Double barrier contraceptives must be used through the trial by both sexes. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test ≤ 72 hours prior to initiating treatment.
20. Liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C). Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. Hepatitis B virus (HBV) DNA and hepatitis C virus (HCV) RNA polymerase chain reaction (PCR) testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.
21. Known diagnosis of human immunodeficiency virus (HIV) infection
22. History of another malignancy within 3 years, except cured basal cell carcinoma of the skin, treated ductal carcinoma in situ (DCIS), cured early stage prostate cancer without detectable prostatic specific antigen (PSA) or excised carcinoma in situ of the cervix
23. Patients should not receive immunization with attenuated live vaccines during study period or within 1 week of study entry. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guérin (BCG), yellow fever, varicella and TY21a typhoid vaccines.
24. Patients taking medications known to be strong CYP3A inhibitors
25. Patients who are currently treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme cytochrome P450, family 3, subfamily A (CYP3A), and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.
26. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
27. Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | During the first cycle of treatment; approximately 4 weeks
  i. Grade 4 hematologic toxicity (excluding anemia) lasting more than 7 days
  ii. Grade 3 anemia lasting more than 7 days or requiring blood transfusion
  iii. Grade 4 anemia
  iv. Grade ≥ 3 febrile neutropenia of any duration
  v. Grade ≥ 3 nausea and or vomiting lasting more than 72 hours in spite of standard supportive therapy
  vi. Grade ≥ 3 non-hematologic toxicity (excluding alopecia)

SECONDARY OUTCOMES:
Clinical benefit rate | During the entire duration of therapy estimated to be an average of 6 months for each patient
  Sum of complete response, partial response and stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Taofeek Owonikoko, MD, PhD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Winship Cancer Institute of Emory University, Atlanta, Georgia, United States

REFERENCES:
- See also: Clinical Trials at Winship — https://winshipcancer.emory.edu/clinical-trials/index.html
- See also: Winship Cancer Institute of Emory University — http://winshipcancer.emory.edu